CLINICAL TRIAL: NCT04174469
Title: First Description of a Severe Ivermectin Neurotoxicity in a Child Carrying ABCB1 Nonsense Mutations.
Brief Title: Ivermectin Neurotoxicity and ABCB1 Gene Mutations
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); INRAE, Toulouse France (Unknown); Université Paris-Saclay, Gif-sur-Yvette, France (Unknown); University Hospital, Montpellier France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0176
Record Dates: First submitted 2019-05-16; First posted 2019-11-22 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-05

CONDITIONS: DNA Sequencing
Keywords: ivermectin; neurotoxicity; ATP binding cassette subfamily B member 1; ABCB1/P-glycoprotein (P-gp); multidrug transporter; drug adverse event; Ivermectin toxicity
MeSH Terms: conditions — Neurotoxicity Syndromes; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample and DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study report a unique case of severe intoxication in a child treated with oral ivermectin to prevent scabies infection. The ABCB1 gene sequencing found the child compound heterozygote for two nonsense mutations, one in each gene copy. The child had inherited from each parent one of the alleles. Each mutation generate a predicted truncated protein that likely lead to ABCB1 loss of function, and the undesirable effects observed.

The study report a unique case of severe intoxication in a child treated with oral ivermectin to prevent scabies infection. The ABCB1 gene sequencing found the child compound heterozygote for two nonsense mutations, one in each gene copy. The child had inherited from each parent one of the alleles. Each mutation generate a predicted truncated protein that likely lead to ABCB1 loss of function, and the undesirable effects observed.

While in some animals, nonsense ABCB1 mutations can lead to neurotoxicity of several ABCB1-substrate drugs, in humans, ivermectin was considered to have an especially high margin of safety, and nonsense mutations have never been reported before, nor has the neurotoxicity of ivermectin apparently caused by these two mutations never been reported before.

This discovery is of critical importance for the child, since it dictates that clinicians would need to optimize any ABCB1 substrate-based therapy in the future. More generally, such information must be brought to the attention of clinicians' medics, and in particular infectious disease specialists, pediatricians, and general practitioners.

It points the importance of pharmacovigilance, and the benefit of pharmacogenomic genotyping in well-defined phenotype, still too rarely considered in clinical practice before the implementation of a drug treatment.

This work results from a multidisciplinary approach, combining several areas of expertise in clinical pediatrics, pharmacology, biology, and bioinformatics.

ELIGIBILITY:
Inclusion Criteria:

* episode of neurotoxicity

Exclusion Criteria:

* NA

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child followed in the pediatric ward of Toulouse University Hospital for the episode of neurotoxicity and his parents
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Patient DNA sequencing | 1 day
  Biological diagnostic: genotyping of ABCB1 (NM_000927.4) by using next generation sequencing (Agilent SureSelectQXT®, Miseq® Illumina). Bio-informatic analysis on JSI medical system GmbH sequence pilot CE v4.3.1 software.
  Identified mutations were subsequently checked using Sanger sequencing on 3130XL (Applied Biosystems®). Bio-informatic analysis on SeqScape v2.5 software.

SECONDARY OUTCOMES:
ivermectin dosage | 1 day
  Biological diagnostic: blood test of ivermectin dosage (normal level: 46,6 (± 21,9) ng/mL for a single dose of 12 mg after 4H; and according to pharmacokinetics informations of VIDAL referential).
cerebral spinal fluid dosages | 1 day
  Cerebrospinal fluid test

CONTACTS AND LOCATIONS:
Overall Officials: Séverine CUNAT, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC